CLINICAL TRIAL: NCT04982887
Title: Comparison of the Effectiveness of Two Different Exercise Programs Adapted to the Tele Rehabilitation Program in Parkinson's Patients During the Covid 19 Pandemic Period
Brief Title: Tele-Rehabilitation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: BElibol (Unknown); NKöse (Unknown); GYÇakmaklı (Unknown)
Responsible Party: Principal Investigator, Emine Nur Demircan, Specialist Physiotherapist / Research Assistant, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tele-Rehabilitation
Record Dates: First submitted 2021-05-09; First posted 2021-07-29 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: Tele Rehabilitation, Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: Exercise
- Control Group (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The cervical region is one of the most affected regions of the musculoskeletal system due to the intensive proprioceptors. Studies have shown that many position sense proprioceptors are over the deep group cervical muscles such as longus colitis and longus capitis. The deep group cervical muscles, which perform a dynamic ligament function, have an important role in maintaining the stability of the spine as well as the proprioceptive sense. In particular, proprioceptive receptors, which are commonly found in the deep suboccipital muscles; There are cervical and reflex connections with vestibular, visual and postural control systems.
  Other Names: Exercise (Servical Stabilization exercises and conventional exercise)

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disease that occurs with the effect of dopaminergic pathways in the substantia nigra and causes a progressive decrease in motor functions. When the literature is examined; Physiotherapy and rehabilitation programs applied in PD include conventional physiotherapy methods and neurophysiological based activity training. Classical physiotherapy programs; It includes stretching, strengthening, aerobics, posture exercises, balance and coordination training. PH treatment in recent years; Virtual reality is gradually enriched with motor imagery and robot-assisted physiotherapy applications and different exercise methods including dance, music therapy, yoga, pilates and spinal stabilization exercises.

Stabilization exercises, which form the basis of spinal stabilization training, use the basic principles of motor learning. The aim of the spinal stabilization exercise program is to support the vertebral column by increasing the strength and endurance of the stabilizer muscles, to improve the spinal posture by increasing kinesthetic awareness and to improve balance control.

The COVID-19 pandemic has highlighted the importance of telerehabilitation practices even more. Telerehabilitation can be defined as providing rehabilitation services remotely using information and communication technologies. In order to minimize the risk of transmission in the COVID-19 pandemic, physical activity levels of individuals have been reduced by restricting social life and the access of sick individuals to rehabilitation services is severely restricted. In addition, rehabilitation professionals are at risk in the treatment of these patients due to the serious transmission risk of COVID-19. Considering these situations, it is emphasized by many authorities that telerehabilitation practices should be expanded.

Inactivity, which occurs as a result of restrictions in access to social isolation and rehabilitation services, brought about by the COVID-19 Pandemic in Parkinson's patients, adversely affects the progression of the disease. Telerehabilitation allows patients who cannot access rehabilitation due to their geographical, economic or physical disabilities to benefit from rehabilitation services. It is known that telerehabilitation applied in various neurological diseases reduces the fatigue levels of the patients, improves their functional activities and quality of life.

In line with all these reasons, this study was planned to investigate the effectiveness of two different exercise programs adapted to the telerehabilitation program in Parkinson's patients during the Covid 19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Parkinson's Disease who came to Hacettepe University between December 2018 and July 2019 were included in the thesis study.
* Individuals who received physiotherapy training two years ago will be contacted by phone and invited to study.
* On these dates, among the individuals selected within the scope of the thesis study, those who agree to participate in the study will be included in the study.

Exclusion Criteria:

-Persons not meeting the above criteria were excluded from the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-08 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | baseline to 6 week after
  Unified Parkinson's Disease Rating Scale. There are 4 sub-parameters. 1. mental status, behavior and mental state 2. daily life activities 3. motor inspection 4. treatment complications. mental status, behavior and mental state total 16 points, daily activity total 52 points, Motor parameter total 92 points, treatment complications total 23 points. Total maximum 183 points. the total score is calculated by adding all sub-parameter scores. low value is good, high value is a symptom of bad result.
Numeric Analog Scale | baseline to 6 week after
  Numerical rating scale of pain intensity. 0 to 10 is a scale with a rating. 0 points no pain 10 points is a scale with very severe pain. The participant is asked to say a value in this range according to the severity of pain.
30 - Second Chair Stand Test | baseline to 6 week after
  It is used to assess individuals' lower extremity strength and static balance. the individual is asked to sit and stand in a chair for 30 seconds.
Static Standing Balance Test | baseline to 6 week after
  Individuals were asked to stand in different positions and their static balance was assessed.
The Fear of Covid-19 Scale | baseline to 6 week after
  It is a test that measures individual's Covid-19 fears. Min:7 Max:35 "high score is bad score."
Short-Form 36 | baseline to 6 week after
  SF-36 (Short Form 36). Quality of life survey. examines 8 dimensions of health with 36 items. physical function, social function, role restrictions, mental health, vitality, pain and general health. The scores of each parameter are between 0 and 100. 0 bad, 100 good results. is calculated by taking the values of the sub-parameters.
Beck Anxiety Inventory | baseline to 6 week after
  Assesses anxiety level. Min:0 Max:63 "high score is bad score."
The Beck Depression Inventory | baseline to 6 week after
  Assesses the level of depression. Min:0 Max: 63 "high score is bad score."
ACTIVLIM Scale | baseline to 6 week after
  It is a questionnaire that measures the activity limitation of individuals. Min: 0 Max:36 "high score is good score."
Standardized Mini Mental Test | baseline to 6 week after
  Evaluates the cognitive level of the person

CONTACTS AND LOCATIONS:
Overall Officials: Ozden BASKAN, Study Director — Istanbul Rumeli University
Locations (1):
- Istanbul Rumeli University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bennett SE, Karnes JL. Neurological Disabilities. Assessment and Treatment. 1 st ed. Lippincott: Philadelphia; 1998.
- [Background] Doherty KM, van de Warrenburg BP, Peralta MC, Silveira-Moriyama L, Azulay JP, Gershanik OS, Bloem BR. Postural deformities in Parkinson's disease. Lancet Neurol. 2011 Jun;10(6):538-49. doi: 10.1016/S1474-4422(11)70067-9. Epub 2011 Apr 22. PMID 21514890
- [Background] Jankovic J. Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):368-76. doi: 10.1136/jnnp.2007.131045. PMID 18344392
- [Background] Vaugoyeau M, Viel S, Amblard B, Azulay JP, Assaiante C. Proprioceptive contribution of postural control as assessed from very slow oscillations of the support in healthy humans. Gait Posture. 2008 Feb;27(2):294-302. doi: 10.1016/j.gaitpost.2007.04.003. Epub 2007 May 16. PMID 17509884
- [Background] Bloem BR, Beckley DJ, van Dijk JG, Zwinderman AH, Remler MP, Roos RA. Influence of dopaminergic medication on automatic postural responses and balance impairment in Parkinson's disease. Mov Disord. 1996 Sep;11(5):509-21. doi: 10.1002/mds.870110506. PMID 8866492